CLINICAL TRIAL: NCT05991713
Title: Individual Differences in Emotional and Behavioral Patterns and Their Relationship to Cognition
Brief Title: Geolocation Positional System (GPS) Experience
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Aaron Heller, Associate Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20150678; R01MH133693 (NIH)
Record Dates: First submitted 2023-08-07; First posted 2023-08-15 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Emotions; Anhedonia; Depression
MeSH Terms: conditions — Anhedonia; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Modifying Exploration (Experimental): Individuals will be asked on certain days to increase their levels of exploration, and some days be asked to decrease their levels of exploration. Participants will do this for up to six months.
  Interventions: Behavioral: Modifying Exploration

INTERVENTIONS:
Behavioral: Modifying Exploration — Participants in this group will use a mobile phone sensor data application that uses an accelerometer, Wireless Fidelity (WiFi) and/or GPS designed for smartphone devices. This technology allows the phones to capture information automatically and passively on the participant's activity. The application will be collecting participants' data 24 hours a day, 7 days a week. Participants will be asked to make alterations to their exploration levels approximately 20 days of their participation in the study.

SUMMARY:
The purpose of this study is to use smartphone technology to capture individual location emotional and cognitive data, to examine how real-world behaviors thoughts, emotions, and brain activity are related to one another.

DETAILED DESCRIPTION:
The observational portion of this study was initially approved in 2015, this is a subset of the initially approved study and it is a clinical trial of 100 participants.

ELIGIBILITY:
Inclusion Criteria:

* Must agree to give informed consent
* Must be willing to have an functional Magnetic Resonance Imaging (FMRI) scan
* Must be able to receive and respond to daily text messages assessing current emotion
* Must be willing to download and run a GPS tracking application (FollowMee) onto their smartphone for a four-month period

Exclusion Criteria:

* history of head trauma, seizures, or neurological disorders
* severe/unstable medical conditions
* conditions that interfere with MRI
* pregnancy
* lifetime psychotic/bipolar disorder
* chronic/severe substance or alcohol abuse/dependence
* antipsychotic medication

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2028-06-15 (Estimated); Study Completion 2028-06-15 (Estimated)

PRIMARY OUTCOMES:
Change in positive emotional response as measured by ecological momentary assessment | Baseline, up to 6 months
  Emotional response will be measured by computing a total mean score of "happy", "excited", "content", "attentive", "relaxed". The total mean score ranges from 0 to 100, with higher scores indicating greater positive emotional response.

SECONDARY OUTCOMES:
Change in negative emotional response as measured by ecological momentary assessment | Baseline, up to 6 months
  Emotional response will be measured by computing a total mean score of "sad", "tired", "upset", "irritable", "anxious". The total mean score ranges from 0 to 100, with higher scores indicating greater negative emotional response.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron S Heller, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No